CLINICAL TRIAL: NCT01183221
Title: The Effects of Oxytocin on Complex Social Cognition in Autism Spectrum Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexander Kolevzon (Other)
Responsible Party: Sponsor-Investigator, Alexander Kolevzon, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: GCO 09-0857
Record Dates: First submitted 2010-08-12; First posted 2010-08-17 (Estimated); Results first posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-03

CONDITIONS: Autism; ASD
MeSH Terms: conditions — Autistic Disorder | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive 24IU intranasal oxytocin or placebo on days separated by a minimum of 3 weeks. Randomization order to drug condition is counter-balanced.
Who Masked: Participant, Investigator
Masking Description: Both the participant and investigator are blind to drug condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Syntocinon then Placebo (Experimental): 24IU intranasal oxytocin, minimum of 3 weeks off, then placebo
  Interventions: Drug: Syntocinon; Drug: Placebo
- Placebo then Syntocinon (Placebo Comparator): Placebo, minimum of 3 weeks off, then 24IU intranasal oxytocin or placebo
  Interventions: Drug: Syntocinon; Drug: Placebo

INTERVENTIONS:
Drug: Syntocinon — One dose of 24 IU (3 sprays/nostril)
  Other Names: Intranasal oxytocin
Drug: Placebo — Intranasal Placebo

SUMMARY:
This study examines the effects of a single dose of intranasal oxytocin (vs. placebo) on complex social cognition in adults with autism spectrum disorders.

DETAILED DESCRIPTION:
Participants receive a one-time administration of 24-IU intranasal oxytocin (or placebo) and perform an empathic accuracy task, a novel and ecologically valid measure of complex social cognition, in conjunction with functional magnetic resonance imaging (fMRI). The investigators will investigate the effects of oxytocin (versus placebo) on the behavioral and neural correlates of empathic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* In good physical health
* Meet criteria for ASD according to psychiatric interview using the Diagnostic and Statistic Manual, Fourth Edition (DSM-IV)
* Must be a history of developmental delay
* Must meet full criteria for ASD on the Autism Diagnostic Interview- Revised (ADI-R) on either the social or communication domains and within two points on other domain (only if parent available for interview)
* Must meet full criteria for ASD on the Autism Diagnostic Observation Schedule- Generic (ADOS-G) on the social domain. Meeting for ASD on the communication domain and total domain is not necessary
* Must have a verbal IQ greater than 75, as measured by the Wechsler Adult Intelligence Scale- Fourth Edition (WAIS- III). Intelligence testing performed at other sites or through another protocol at this site within the past year will also be accepted
* Capability of performing experimental tasks (i.e. can read and understand task instructions, cooperate with procedures)
* Informed consent and capacity
* Female participants must remain on birth control for the duration of the study

Exclusion Criteria:

* Participants with any primary psychiatric diagnosis at screening
* Participants with a medical history of neurological disease, including, but not limited to, epilepsy/seizure disorder (except simple febrile seizures), movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes, or known abnormal MRI/structural lesion of the brain
* Participants who are pregnant, who gave birth in the last six months, or who are currently breastfeeding
* Participants with a medical condition that might interfere with the conduct of the study, confound interpretation of the study results, or endanger their own well-being
* Participants with evidence or history of malignancy or any significant hematological endocrine, cardiovascular (including rhythm disorder), respiratory, renal, hepatic, gastrointestinal disease, or other major medical conditions
* Participants taking psychoactive medication(s) (e.g., stimulants, antidepressants, antipsychotics, antiepileptics, anxiolytics, clondine)
* Participants who, in the Investigator's opinion, might not be suitable for the study
* Participants who are involved in another study whose procedures could influence performance in the current study
* Female participants who do not stay on birth control for the duration of the study
* Participants who have a known contraindication to the MRI scan: including sever claustrophobia or any kind of metal implant in the body

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06-18 (Actual); Primary Completion 2014-04-25 (Actual); Study Completion 2014-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Bartz, P.h.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine - Seaver Autism Center for Research and Treatment, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Syntocinon Then Placebo: One dose 24IU (3 sprays/nostril) intranasal oxytocin, minimum of 3 weeks off, then Intranasal placebo
- Placebo Then Syntocinon: Intranasal Placebo, minimum of 3 weeks off, then 24IU (3 sprays/nostril) intranasal Syntocinon
Period: First Dose
Arm/Group | Syntocinon Then Placebo | Placebo Then Syntocinon
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: 3 Weeks Wash Out
Arm/Group | Syntocinon Then Placebo | Placebo Then Syntocinon
Started | 15 | 15
Completed | 14 | 14
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Second Dose
Arm/Group | Syntocinon Then Placebo | Placebo Then Syntocinon
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Syntocinon Then Placebo | Placebo Then Syntocinon | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (8.9) | 27.5 (6.7) | 29.3 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Empathic Accuracy Performance
Description: Participants watch videos of targets describing positive and negative autobiographical events and provide continuous ratings of how positive-negative the target is feeling on a 9-point Likert scale. Empathic accuracy is operationalized as a timecourse correlation between perceiver inferences about target affect and targets' own affect ratings.
Time Frame: 45 minutes after drug/placebo administration
Population: The computer in the imaging suite crashed and the behavioral outcome data were not adequately backed up. The imaging data cannot be analyzed while pts were performing the EA task because without the behavioral data, the researchers do not know what pts were doing at each timepoint (it was an event related design). The researchers would not have the necessary information to know how to segment the data or what trial type (self/other/control) pts were doing at the various time points.
Arm/Group | Syntocinon Then Placebo | Placebo Then Syntocinon
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Fmri BOLD Response During Empathic Accuracy Task
Description: Images will be acquired using a 3.0 Tesla Siemens Allegra MRI scanner equipped to acquire gradient-echo, echoplanar T2*-weighted images (EPI) with blood oxygenation level dependent (BOLD) contrast. Each volume will comprise 26 axial slices of 4.5mm thickness and a 3.5 x 3.5mm in-plane resolution, aligned along the AC-PC axis. Volumes will be acquired continuously every 2 seconds. Each run will begin with 5 'dummy' volumes, which will be discarded from further analyses. At the end of the scanning session, a T-1 weighted structural image will be acquired from each participant.
Time Frame: 45 minutes after oxytocin/placebo administration
Population: as for outcome 1
Arm/Group | Syntocinon Then Placebo | Placebo Then Syntocinon
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Syntocinon: One dose 24IU (3 sprays/nostril) intranasal oxytocin,
Arm/Group | Syntocinon | Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 8/28 | 10/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Syntocinon (N=28) | Placebo (N=28)
Ringing Ears (Ear and labyrinth disorders) | 0 | 1
Headache (General disorders) | 4 | 2
Fatigue (General disorders) | 2 | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Watery eyes (Endocrine disorders) | 1 | 2
Sore throat (Skin and subcutaneous tissue disorders) | 0 | 1
Cold hand (Skin and subcutaneous tissue disorders) | 0 | 1
Dizzy (General disorders) | 0 | 1 — when got up from fMRI scan table
Burning in throat after nasal spray (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sinuses tender (Blood and lymphatic system disorders) | 2 | 0
Lack of focus (Psychiatric disorders) | 1 | 2
Felt body/joint pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Breasts tender (Reproductive system and breast disorders) | 1 | 0
Difficulty sleeping (Psychiatric disorders) | 1 | 0
Light headedness (General disorders) | 0 | 1
Slowed thought process (Psychiatric disorders) | 1 | 0
Runny nose (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Difficulty hearing (Ear and labyrinth disorders) | 1 | 1
Chest tightness (Cardiac disorders) | 0 | 1 — vital signs stable
Mild diarrhea (Gastrointestinal disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes